CLINICAL TRIAL: NCT02053805
Title: Personalized Prostate Cancer Screening Among Men With High Risk Genetic Predisposition- a Prospective Cohort Study
Brief Title: Prostate Cancer Screening Among Men With High Risk Genetic Predisposition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0582_13_RMC
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: BRCA1 Syndrome; BRCA2 Syndrome; Lynch Syndrome
Keywords: prostate cancer; BRCA1 Syndrome; BRCA germ-line mutation; Lynch syndrome; BRCA2 Syndrome
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- screening tests (Other): The screening will include: DRE, PSA , a multiparametric prostate MRI and a trans-rectal ultra-sound guided prostate biopsy/ MRI-US fusion , IPSS questionnaire, trans-rectal US assessment of prostate size, urine flow and residual.
  Interventions: Other: PSA; Other: IPSS questionnaire; Other: DRE (Digital Rectal Examination ); Other: urine flow and residual; Procedure: a multiparametric prostate MRI; Procedure: trans-rectal ultra-sound guided prostate biopsy

INTERVENTIONS:
Other: PSA — PSA. Serum & plasma will be stored for future investigations
Other: IPSS questionnaire — the validated International Prostate Symptom Score
Other: DRE (Digital Rectal Examination ) — physical examination for the prostate gland
Other: urine flow and residual — The post void residual will be recorded by using ultrasound. Creatinine level will be checked.
Procedure: a multiparametric prostate MRI — The MRI will be reported on a 5 point Likert Scale
Procedure: trans-rectal ultra-sound guided prostate biopsy — 12 core Trans-rectal prostatic biopsy for diagnostic purposes

SUMMARY:
This will be a prospective diagnostic trial of screening for prostate cancer among men with genetic predisposition.

DETAILED DESCRIPTION:
This will be a prospective diagnostic trial of screening for prostate cancer among men with genetic predisposition. The target population is males (40-70 year old) carrying a BRCA1 and/or BRCA2 germ line mutation. They will be identified via our Genetic counseling unit. All men after signing an informed consent will undergo the following tests: PSA, free to total PSA, MRI of prostate and prostate biopsy. The primary endpoint will be to estimate the prevalence, stage and grade of prostate cancer in this population. Additionally, the study aims to estimate the impact of these germ line mutations on benign prostatic hyperplasia. Furthermore, this study aims to create a bio-bank of tissue, urine and serum of this unique cohort for future investigations. Finally, this study will identify an inception cohort for future interventional studies of primary and secondary prevention.

ELIGIBILITY:
Inclusion Criteria:

* Male carrier of mutation in BRCA 1\2 or germ-line mutations in the MMR genes (MLH1, MSH2 , MSH6 or PMS2).
* WHO performance status 0-2 (Appendix 2)
* Absence of any psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow-up schedule.
* Individuals that cannot undergo the MRI exam due to high creatinine level or claustrophobic will be disc loud from the MRI part.
* Informed written consent must be sought according to ICH/EU GCP, before subject registration.

Exclusion Criteria:

* Previous cancer with a terminal prognosis of less than five years.
* Previous prostate cancer

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence, stage and pathology of screen-detected prostate cancer in BRCA1/BRCA2 founder mutation carriers and Lynch mutation carriers | within 2 years

SECONDARY OUTCOMES:
Accuracy of different screening tests (PSA, free to total PSA, prostate MRI) in detecting prostate cancer among men with genetic predispositions. | within 2 years

OTHER OUTCOMES:
Accuracy of different screening tests (PSA, free to total PSA, prostate MRI) in detecting clinically significant prostate cancer among men with genetic predispositions. | within 2 years
Cost effectiveness of different screening tests (PSA, free to total PSA, prostate MRI) in detecting prostate cancer and clinically significant prostate cancer among men with genetic predispositions. | within 2 years
Impact of genetic mutations (BRCA, Lynch) on lower urinary tract symptoms (IPSS, flow and post void urine residual) and BPH ( benign prostatic hyperplasia). | within 2 years
Genomic and biological profiles in samples from BRCA and Lynch mutation carriers and characterize changes related to prostate cancer. | within 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Margel, MD PhD, Principal Investigator — Rabn Medical Center, Beilinson Campus
Locations (2):
- Israel (2):
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Segal N, Ber Y, Benjaminov O, Tamir S, Yakimov M, Kedar I, Rosenbaum E, Sela S, Ozalvo R, Shavit-Grievink L, Keder D, Baniel J, Margel D. Imaging-based prostate cancer screening among BRCA mutation carriers-results from the first round of screening. Ann Oncol. 2020 Nov;31(11):1545-1552. doi: 10.1016/j.annonc.2020.06.025. Epub 2020 Sep 18. PMID 32958357
- [Derived] Margel D, Benjaminov O, Ozalvo R, Shavit Grievink L, Kedar I, Yerushalmi R, Ben-Aharon I, Neiman V, Yossepowitch O, Kedar D, Levy Z, Shohat M, Brenner B, Baniel J, Rosenbaum E. Personalized prostate cancer screening among men with high risk genetic predisposition- study protocol for a prospective cohort study. BMC Cancer. 2014 Jul 21;14:528. doi: 10.1186/1471-2407-14-528. PMID 25047061